CLINICAL TRIAL: NCT03380728
Title: Tolerability and Efficacy of Ibogaine in the Treatment of Alcoholism: an Open-label Escalating-dose Trial
Brief Title: Ibogaine in the Treatment of Alcoholism: an Open-label Escalating-dose Trial
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Sao Paulo (Other)
Collaborators: Coordenação de Aperfeiçoamento de Pessoal de Nível Superior. (Other Government); Conselho Nacional de Desenvolvimento Científico e Tecnológico (Other Government); International Center for Ethnobotanical Education, Research, and Service (Other)
Responsible Party: Principal Investigator, Rafael Guimarães dos Santos, Postdoctoral Fellow, Principal Investigator, University of Sao Paulo
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 72938717.3.0000.5440
Record Dates: First submitted 2017-12-15; First posted 2017-12-21 (Actual); Last update posted 2024-11-26 (Actual); Status verified 2024-11

CONDITIONS: Alcoholism
MeSH Terms: conditions — Alcoholism

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Ibogaine (Experimental): Ibogaine Hydrochloride 240 mg on day 1, placebo on day 4, placebo on day 7
  Interventions: Drug: Ibogaine Hydrochloride

INTERVENTIONS:
Drug: Ibogaine Hydrochloride — The first 3 patients will receive oral doses of 20 to 400 mg of ibogaine in an open-label design. If the 3 higher doses (240, 320 and 400 mg) are well tolerated, the next 9 volunteers will receive these doses or placebo randomly in 3 different groups.
  Other Names: Placebo

SUMMARY:
Approximately 5% of the world's adult population has some alcohol-related disorder, which in addition is associated with 3% of all deaths in the world. In Brazil, harmful use and dependence on alcohol reach about 10% of the population, with alcohol being one of the main factors of disease and mortality. Although the medications currently used have some efficacy, the adverse effects and relatively long time of treatment are factors that may reduce patients' motivation to continue taking the medication correctly. Therefore, it is necessary to conduct research with new drugs for the treatment of alcoholism. Ibogaine is an alkaloid present in the bush Tabernanthe iboga (iboga), a plant from Central Africa traditionally used in countries such as Gabon and Cameroon. Animal studies and case series suggest that one or a few doses of ibogaine significantly reduce withdrawal symptoms and the intensity of use of various drugs, including opioids, psychostimulants, and alcohol. However, there are no controlled clinical studies that have explored these effects. The aim of the present study is to evaluate the safety, tolerability and efficacy of increasing doses of ibogaine in 12 alcoholic patients. Each patient will be hospitalized for 20 days and receive 3 increasing doses of ibogaine. The first 3 patients will receive oral doses of 20 to 400 mg of ibogaine in an open-label design. If the 3 higher doses (240, 320 and 400 mg) are well tolerated, the next 9 volunteers will receive these doses or placebo randomly. The volunteers will also be evaluated 7, 14 and 21 days and 1, 3, 6 and 12 months after leaving the hospital to monitor the consumption of alcohol and other drugs.

ELIGIBILITY:
Inclusion Criteria:

* Literate people
* Diagnosis of alcoholism assessed by the Structured Clinical Interview for Diagnostic and Statistical Manual of Mental Disorders (SCID-V)
* History of at least two previous failed treatments for alcoholism (with drug use and / or psychotherapy)
* Signing the Free and Informed Consent Form.

Exclusion Criteria:

* Presence of any psychiatric diagnosis (excluding alcohol / tobacco / nicotine abuse / dependence) assessed by the SCID-V
* Presence of clinical disease (especially cardiovascular and hepatic diseases), based on interview, physical and laboratory examination (hemogram and electrocardiogram, ECG)
* Absence of family or personal history of bipolar disorder and psychotic disorders
* Absence of recent symptoms of hypomania, mania or psychosis
* Non-literate people
* Pregnant or lactating women
* Recent use of illicit drugs (confirmed by examination in urine).

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2022-10-30 (Actual); Primary Completion 2024-10-30 (Actual); Study Completion 2024-10-30 (Actual)

PRIMARY OUTCOMES:
Time without using alcohol | 0-1 month
  Daily alcohol use

SECONDARY OUTCOMES:
Subjective effects | 0-12 hours
  Acute and subacute subjective effects
Cardiovascular effects | 0-72 hours
  Electrocardiogram

CONTACTS AND LOCATIONS:
Overall Officials: Rafael dos Santos, PhD, Principal Investigator — Departamento de Neurociências e Ciências do Comportamento, Faculdade de Medicina de Ribeirão Preto, Universidade de São Paulo; Jaime Hallak, PhD, Study Director — Departamento de Neurociências e Ciências do Comportamento, Faculdade de Medicina de Ribeirão Preto, Universidade de São Paulo
Locations (1):
- Ribeirão Preto Medical School, Ribeirão Preto, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: dos Santos RG, Bouso JC, Hallak JEC. The antiaddictive effects of ibogaine: A systematic literature review of human studies. Journal of Psychedelic Studies 1(1): 20-28, 2017. — http://akademiai.com/doi/abs/10.1556/2054.01.2016.001
- See also: Clare W et al. Detoxification from methadone using low, repeated, and increasing doses of ibogaine: A case report. Journal of Psychedelic Studies 1(1): 29-34. — http://akademiai.com/doi/abs/10.1556/2054.01.2017.005